CLINICAL TRIAL: NCT03314571
Title: Obstetrical Analgesia in the Estaing Hospital Maternity. A Prospective Database to Study the Determinants of Labor Pain and the Resulting Maternal Non Satisfaction.
Acronym: AOMHE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-357; 2017-A00814-49 (Other: 2017-A00814-49)
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Epidural Analgesia; Hospital Follow-up
Keywords: Epidural analgesia; Labor pain; Satisfaction; Care assessment; Psychometry
MeSH Terms: conditions — Labor Pain; Personal Satisfaction | interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non applicable
  Interventions: Other: analgesia for labor

INTERVENTIONS:
Other: analgesia for labor — A prospective database to study the determinants of labor pain and the resulting maternal non satisfaction.

SUMMARY:
There is a trend to offer personalized care in many medical domains. In the field of labor pain, it appears that maternal satisfaction about care is multifactorial, and that labor pain is only one of its determinants, competing with psychological and sociological factors. Furthermore, labor pain is also multifactorial, depending on predisposition to pain, the way analgesia is conducted, and other environmental factors. We wish to develop predicting models of maternal satisfaction, in order to offer in the future a better tailored analgesia.

DETAILED DESCRIPTION:
The observation shall be conducted at 3 major points of measurement throughout labor:

1. Pre-, i.e. at the systematic visit for anesthesia, during the 3rd trimester of pregnancy. The collected variables will be: demographic, morphometric, socioeconomic, psychometric. The latter shall consist in a short questionnaire-based assessment by: Hospital Anxiety and Depression Scale, 5-points Mental Health Inventory, Life Orientation Scale. As soon as it will be validated, a Pain Sensitivity Questionnaire shall be added.
2. Intra-, i.e. clinical data from the anesthesia file: conduction of epidural analgesia, labor pain, drug consumption, obstetrical outcomes.
3. Post-, i.e. maternal satisfaction assessed by a set of seven 11-point numerical rating scales at day2 post childbirth, along with a written short qualitative assessment.

Different multivariable statistical models shall be used to identify the patients profiles and the possible determinants of satisfaction: descriptive (factorial analyses) and inferential (GLM or longitudinal).

ELIGIBILITY:
Inclusion Criteria:

* Any parturient coming for her regular pre-partum anesthesia visit at the Estaing Hospital Maternity

Exclusion Criteria:

* Refusal of epidural analgesia at the time of the visit.
* Participation refusal.
* Inability to answer the pre- or post-partum questionnaires.
* Any medical condition considered as a relevant exclusion criterion by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal satisfaction about analgesia for labor | from the morning of day 2 postpartum to the morning of day 3 postpartum.
  Eight-domain questionnaire designed for the purpose of the study, each domain being addressed by an 11-point numerical scale from 0 (not satisfied at all) to 10 (totally satisfied). The 8 domains are: general analgesia care, rapidity of analgesia, pain control at expulsion, mobility during labor, self-control of labor, caregivers' attention, pain at epidural puncture, information about epidural.

SECONDARY OUTCOMES:
Wish for a similar analgesia for future labor. | from the morning of day 2 postpartum to the morning of day 3 postpartum.
Qualitative maternal concerns about analgesia for labor | from the morning of day 2 postpartum to the morning of day 3 postpartum
  verbatim (free field).

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte STORME, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France